CLINICAL TRIAL: NCT01405183
Title: Association Between Hepatitis C Infection and Renal Cell Carcinoma, a Case Control Study
Brief Title: Association Between Hepatitis C Infection and Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Principal Investigator, Humberto C. Gonzalez, MD, Henry Ford Health System
Other Study IDs: P08406
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hepatitis C; Renal Cell Carcinoma; Colorectal Cancer
Keywords: Hepatitis C; Renal Cell Carcinoma; Colorectal Cancer
MeSH Terms: conditions — Hepatitis C; Carcinoma, Renal Cell; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hepatits C antibody Hepatitis C RNA quantitative Hepatitis C Genotype
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Renal Cell Carcinoma patients: Newly diagnosed (within 6 months) renal cell carcinoma patients in who a biopsy or surgery will be performed
  Interventions: Other: Hepatitis C testing
- Colorectal cancer patients: Newly diagnosed (6 months) colon cancer patients
  Interventions: Other: Hepatitis C testing

INTERVENTIONS:
Other: Hepatitis C testing — Hepatitis C antibody, Hepatitis C RNA quantitative and for those who test positive Hepatitis C genotype

SUMMARY:
The purpose of this study is to determine if there is an association between hepatitis C infection and kidney cancer. All patients who are diagnosed with kidney cancer and who will either have a biopsy or surgery will be offered to be tested for hepatitis C. The control group will be colon cancer patients. Both groups would be of recent diagnosis (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years or older in whom renal cell carcinoma is suspected and are scheduled for either biopsy or partial or total nephrectomy. Diagnosis within 6 months.
* Male and female patients 18 years or older in whom colorectal cancer has been diagnosed within the last 6 months

Exclusion Criteria:

* Patients who are unwilling to provide consent
* Patients who decline to complete a questionnaire
* Patient in who blood sample cannot be obtained
* Diagnosis of renal cell carcinoma or colon cancer greater than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal cell carcinoma patients will be identified from the urology clinic and from the hospital wards.
  Colorectal cancer patient will be identifed from the hospital wards, pathology reports and gastroenterology endoscopy suits.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2011-01; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of hepatitis C in renal cell carcinoma patients | 2 years
  Determine the prevalence of hepatitis C infection in newly diagnosed renal cell carcinoma patients

CONTACTS AND LOCATIONS:
Overall Officials: Humberto C Gonzalez, MD, Principal Investigator — Henry Ford Hospital; Stuart C Gordon, MD, Study Chair — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Background] Gordon SC, Moonka D, Brown KA, Rogers C, Huang MA, Bhatt N, Lamerato L. Risk for renal cell carcinoma in chronic hepatitis C infection. Cancer Epidemiol Biomarkers Prev. 2010 Apr;19(4):1066-73. doi: 10.1158/1055-9965.EPI-09-1275. Epub 2010 Mar 23. PMID 20332260